CLINICAL TRIAL: NCT03093051
Title: A Clinical Feasibility Study to Evaluate the Safety and Performance of Low-Energy Unpinning Termination Therapy in Patients With VT
Brief Title: Unpinning Termination Therapy for VT (US)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor ceased operations
Sponsor: Cardialen, Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CL005; 2R44HL107055-02 (NIH)
Record Dates: First submitted 2017-03-13; First posted 2017-03-28 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Ventricular Tachycardia
Keywords: Termination; Unpinning; Therapy
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Intervention Model Description: Patients undergoing a routine clinically indicated procedure will have the investigational therapy delivered during the clinically indicated procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- UPT Treatment (Experimental): Investigational therapy (UPT)
  Interventions: Device: Unpinning Termination therapy

INTERVENTIONS:
Device: Unpinning Termination therapy — Electrotherapy comprised of standard biphasic and monophasic pacing pulses
  Other Names: Multi-Stage Therapy; Multi-Stage Electrotherapy

SUMMARY:
This observation study evaluates the safety and performance of UPT therapy in subjects during either an indicated ventricular tachycardia ablation procedure or an ICD implant procedure.

DETAILED DESCRIPTION:
This non-blinded, single-arm open-label, phase 1 pilot, acute research feasibility trial aims to demonstrate that the safety and effectiveness of Unpinning Termination (UPT) electrotherapy observed in the canine can be translated to humans and to demonstrate the safety and performance of UPT electrotherapy in the human population most likely to benefit from this therapy. This study evaluates the safety and performance of UPT therapy in subjects during either an indicated ventricular tachycardia (VT) catheter ablation or an indicated initial implant or device replacement of an implantable cardioverter defibrillator (ICD).

ELIGIBILITY:
Inclusion Criteria:

The subject must meet all of the following inclusion criteria:

1. Life expectancy of 1 year or greater
2. Male or female between 18 and 80 years of age
3. Willing and able to comply with the study protocol, provide a written informed consent
4. Indication for an endocardial VT catheter ablation for symptomatic VT with use of CESS V1.0 or CESS V1.1 OR an indication for an ICD procedure (de novo implant, replacement or upgrade) or de novo CRTD procedure for the risk of or presence of VT (CESS 1.0 and 1.1)
5. Etiology of arrhythmia, or risk of arrhythmia being ischemic cardiomyopathy or non-ischemic cardiomyopathy
6. Medically stable at time of consent to undergo DFT testing performed under general anesthesia or conscious sedation as determined by the investigator

Exclusion Criteria:

The subject must not meet any of the following exclusion criteria:

1. Medically unstable at time of study and unsafe to undergo DFT testing under general anesthesia or conscious sedation as determined by the investigator
2. Hemodynamic instability as determined by the investigator
3. AF or atrial flutter at time of Study Procedure and no anticoagulation for preceding 3 weeks and no preoperative transesophageal echocardiographic, Cardiac CT or Intracardiac echocardiographic confirmation of the absence of LA thrombus
4. Presence of intracardiac thrombus
5. Inability to pass catheters to heart due to vascular limitations
6. Cardiovascular anatomical defects that would complicate placement of the lead or catheter required by the protocol, including congenital heart disease and cardiac vein anomalies as determined by the investigator
7. Pregnancy confirmed by test within 7 days of procedure
8. Presence of a chronically implanted lead in the CS
9. Presence of a ventricular assist device, including intra-aortic balloon pump
10. Subjects indicated for VT ablation and experiencing VF
11. Subjects requiring the use of inotropes and/or vasopressors for hemodynamic support within the 3 days prior to the study
12. Prior VT catheter ablation with associated hemodynamic compromise despite pressor agents or stroke
13. Incessant VT/VF or VT/VF storm within six months of scheduled procedure
14. LVEF < 20%
15. New York Heart Association (NYHA) Class IV heart failure
16. Planned epicardial VT ablation on the same day as the research study
17. History of hyper-coagulable state that could increase risk of thromboembolic events
18. History of hemodynamic compromise due to valvular heart disease requiring IV inotropes or other circulatory support
19. Unstable coronary artery disease as determined by the investigator
20. Severe proximal three-vessel or left main coronary artery disease, without revascularization as determined by the investigators
21. History of embolic stroke, Transient Ischemic Attack or other thromboembolic event in the past 6 months
22. History of Hypertrophic Cardiomyopathy, Arrhythmogenic Right Ventricular Dysplasia, Congenital Heart Anomaly, Cardiac Amyloidosis, Genetic Cardiac Channelopathy or Cardiac Sarcoidosis
23. Cardiovascular surgery or intervention within 1 month prior to enrollment or planned for up to 1 month after enrollment (other than the planned treatment procedure)
24. Morbid obesity: BMI>39 kg/m2
25. Cognitive or mental health status that would interfere with study participation and proper informed consent
26. Presence of mechanical tricuspid valve
27. Active Endocarditis
28. Ventricular arrhythmia with etiology of sarcoid flare
29. Previously implanted lead is under recall by manufacturer or evidence of lead failure as determined by the investigator
30. End Stage Renal Disease on hemodialysis or peritoneal dialysis, or creatinine clearance <15 ml/min
31. Any other medical condition which may affect the outcome of this study or safety of the subject as determined by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Arrhythmia Termination as assessed by the number of episodes restored to sinus rhythm | During study procedure
  Assess the safety and performance of the Cardialen External Stimulation System and safety and performance ofUPT therapy

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H. Cooper, MD, Principal Investigator — Washington University School of Medicine
Locations (7):
- United States (7):
  - Mercy Medical Group, Sacramento, California
  - MercyOne Des Moines Medical Center, Des Moines, Iowa
  - Minneapolis VA Healthcare System, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - OhioHealth Riverside Methodist Hospital, Columbus, Ohio
  - Baylor Scott & White Heart and Vascular Hospital, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Janardhan AH, Gutbrod SR, Li W, Lang D, Schuessler RB, Efimov IR. Multistage electrotherapy delivered through chronically-implanted leads terminates atrial fibrillation with lower energy than a single biphasic shock. J Am Coll Cardiol. 2014 Jan 7-14;63(1):40-8. doi: 10.1016/j.jacc.2013.07.098. Epub 2013 Sep 26. PMID 24076284
- [Background] Janardhan AH, Li W, Fedorov VV, Yeung M, Wallendorf MJ, Schuessler RB, Efimov IR. A novel low-energy electrotherapy that terminates ventricular tachycardia with lower energy than a biphasic shock when antitachycardia pacing fails. J Am Coll Cardiol. 2012 Dec 11;60(23):2393-8. doi: 10.1016/j.jacc.2012.08.1001. Epub 2012 Nov 7. PMID 23141483
- [Background] Li W, Janardhan AH, Fedorov VV, Sha Q, Schuessler RB, Efimov IR. Low-energy multistage atrial defibrillation therapy terminates atrial fibrillation with less energy than a single shock. Circ Arrhythm Electrophysiol. 2011 Dec;4(6):917-25. doi: 10.1161/CIRCEP.111.965830. Epub 2011 Oct 6. PMID 21980076
- [Background] Efimov I, Ripplinger CM. Virtual electrode hypothesis of defibrillation. Heart Rhythm. 2006 Sep;3(9):1100-2. doi: 10.1016/j.hrthm.2006.03.005. Epub 2006 Mar 10. No abstract available. PMID 16945810
- [Background] Ripplinger CM, Krinsky VI, Nikolski VP, Efimov IR. Mechanisms of unpinning and termination of ventricular tachycardia. Am J Physiol Heart Circ Physiol. 2006 Jul;291(1):H184-92. doi: 10.1152/ajpheart.01300.2005. Epub 2006 Feb 24. PMID 16501014
- [Background] Li W, Ripplinger CM, Lou Q, Efimov IR. Multiple monophasic shocks improve electrotherapy of ventricular tachycardia in a rabbit model of chronic infarction. Heart Rhythm. 2009 Jul;6(7):1020-7. doi: 10.1016/j.hrthm.2009.03.015. Epub 2009 Mar 11. PMID 19560090
- [Background] Ambrosi CM, Ripplinger CM, Efimov IR, Fedorov VV. Termination of sustained atrial flutter and fibrillation using low-voltage multiple-shock therapy. Heart Rhythm. 2011 Jan;8(1):101-8. doi: 10.1016/j.hrthm.2010.10.018. Epub 2010 Oct 19. PMID 20969974